CLINICAL TRIAL: NCT03458598
Title: Measuring the Analgesic Effect of Adding Pre-Operative Single Shot Rectus Sheath Blocks to Post-Operative Rectus Sheath Continuous Blocks for Major Urologic Surgery: A Randomized Controlled Trial
Brief Title: Pre-Operative Single Shot Rectus Sheath Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00078459
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Bladder Neoplasm; Prostate Neoplasm; Pelvic Neoplasm; Urologic Neoplasms; Opioid Use; Anesthesia, Local; Pain, Postoperative
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Pelvic Neoplasms; Urologic Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The intra-operative anesthesiologist, surgeon and outcomes assessor are blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single shot rectus sheath block (Experimental): The treatment group will have pre-operative ultrasound-guided single shot bilateral rectus sheath blocks with 20 ml of a ropivacaine / bupivacaine mixture per side.
  Interventions: Procedure: Rectus sheath block; Procedure: Bilateral rectus sheath catheter; Drug: Patient controlled opioid analgesia (PCA)
- Placebo Control (Sham Comparator): The control group will have a pre-operative sham ultrasound-guided subcutaneous injection of 1ml saline per side.
  Interventions: Procedure: Bilateral rectus sheath catheter; Drug: Patient controlled opioid analgesia (PCA); Procedure: Subcutaneous injection saline placebo

INTERVENTIONS:
Procedure: Rectus sheath block — Rectus sheath block under ultrasound
  Arms: Single shot rectus sheath block
Procedure: Bilateral rectus sheath catheter — A nerve block catheter known as a continuous rectus sheath block is inserted by the surgeon at the end of the operation. An infusion of 0.2% ropivacaine is delivered through this for up to 48 hours post-operatively.
Drug: Patient controlled opioid analgesia (PCA) — Patients in both groups will have PCA dilaudid or morphine prescribed for the post-operative period.
Procedure: Subcutaneous injection saline placebo — Subcutaneous injection of 1ml of normal saline under ultrasound guidance at the same site bilaterally as rectus sheath blockade is performed
  Arms: Placebo Control

SUMMARY:
Objectives The primary objective is to demonstrate that in patients undergoing major urologic surgery, Patient Controlled Analgesia (PCA) opioid consumption in the first 24 hours after surgery will be significantly less in patients who have had a single shot rectus sheath block pre-operatively in addition to a post-operative rectus sheath continuous block via surgically placed catheter versus those who only have post-operative rectus sheath continuous block. Secondary outcomes will be opioid requirement intra-operatively, Numerical Rating Scale (NRS) pain scores including maximum pain score in Post Anesthesia Care Unit (PACU) and score at 24 and 48 hours, incidence and severity of nausea, number of vomiting episodes, sedation score, time to first bowel movement, time to first mobilization and duration of hospital stay.

DETAILED DESCRIPTION:
Purpose: To improve analgesia and reduce opioid consumption in patients undergoing major urologic surgery.

Hypothesis: Patients receiving pre-operative single shot rectus sheath blockade in addition to continuous rectus sheath catheters will use less PCA opioid in the first 24 hours post-operatively compared to patients receiving continuous rectus sheath blockade for major urologic surgery.

Justification:

The sensorimotor innervation of the anterior abdominal wall is supplied by the ventral rami of the thoracolumbar spinal (T7-L1) segmental nerves. The thoracolumbar nerves course along the anterolateral wall within the transversus abdominis plane (TAP), and continue anteromedially, before entering the lateral aspect of the posterior rectus sheath. The nerves provide both muscular and cutaneous branches to innervate the muscle fibers and overlying skin with innervation from both left and right nerves supplying the midline. Regional anesthesia techniques for the anterior abdominal wall include both TAP and rectus sheath blocks.

The TAP block has been investigated extensively and shown to reduce opioid analgesia requirements post-operatively. The main difference between TAP block and rectus sheath block is that the rectus sheath block targets the nerves at a more anterior location. Bilateral rectus sheath nerve blocks are required to provide cover for midline incision and the investigators have previously described rectus sheath block with nerve catheter insertion under ultrasound guidance for midline laparotomy. A recent retrospective review from Dutton et al on the use of rectus sheath catheters for major urologic surgery reported that they offer an effective and safe method of peri-operative analgesia in patients undergoing major open urological pelvic surgery. Tudor et al demonstrated that rectus sheath catheters provide analgesia equivalent to that provided by epidurals following laparotomy for colorectal surgery.

At the University of Alberta Hospital, patients having major urologic surgery e.g. cystectomy have surgically placed rectus sheath catheters sited at the end of the procedure as a standard of analgesia care. This is combined with patient-controlled analgesia (PCA) opioid as part of a multimodal approach to post-operative pain control.

One disadvantage of surgically placed TAP and rectus sheath catheters is that they are inserted at the end of surgery. Therefore, the patient does not benefit from them intra-operatively and other methods of analgesia including opiates are required to reduce the sympathetic response to surgical stimulation and to prevent excessive immediate and early post-operative pain. The surgically placed rectus sheath catheters are sited during wound closure and then bolused with local anesthetic just prior to emergence so often the block is not fully established in the early post-operative period resulting in further opiate analgesia requirement.

The primary objective is to demonstrate that in patients undergoing major urologic surgery PCA opioid consumption in the first 24 hours after surgery will be significantly less in patients who have had an ultrasound-guided single shot rectus sheath block pre-operatively in addition to a post-operative rectus sheath continuous block via surgically placed catheter versus those who only have post-operative rectus sheath continuous block.

Secondary outcomes will be opiate requirement intra-operatively, Numerical Rating Scale (NRS) pain scores including pain score in PACU and score at 24 and 48 hours, incidence and severity of nausea, number of vomiting episodes, sedation scores, time to first bowel movement, time to first mobilization and duration of hospital stay.

Research Methods: A randomized, double-blinded controlled trial.

Subjects who meet eligibility criteria will be invited to participate in the study by the clinical care team or research assistant in the Preadmission Clinic. Informed consent will be obtained by the research assistant. Next, all eligible participants will be randomized to the treatment group i.e. pre-operative single shot bilateral rectus sheath blocks + post-operative catheters or the control group i.e. post-operative catheters.

Randomization will be conducted through stratified-blocked randomization with varying blocks of 4 to 6 according to a schedule not known to the investigators using a computerized algorithm. The patient, intra-operative anesthetist, the surgeon and the assessor will be blinded to the randomization assignment.

The treatment group will have pre-operative single shot bilateral rectus blocks with 20 ml of a ropivacaine / bupivacaine mixture per side. The control group will have a pre-operative sham subcutaneous injection of 1ml saline per side. Both groups will have bilateral rectus sheath catheters placed surgically at the end of the procedure. Under direct visualization, the surgeon will insert a standard nerve block catheter between the rectus abdominis muscle and the posterior rectus sheath lateral to the incision on both sides. The catheter will be fixed to skin via a specialized taping system. An infusion of 0.2% ropivacaine will be administered through the rectus sheath catheter (1ml / hour continuous infusion with 15 ml /hour bolus every 4 hours). All patients will receive an IV morphine or dilaudid PCA and adjunctive post-operative medication. Intra-operative morphine / dilaudid administered intra-operatively will be recorded as well as total morphine / dilaudid used in the first 24 hours. Anesthesia technique will be standardized for short-acting opioid use i.e. fentanyl. Peri-operative multimodal analgesia adjuncts will include ketamine 0.2mg/kg and dexamethasone 6mg. All patients will be pre-medicated with acetaminophen 1g and gabapentin 300mg pre-operatively.

Primary and secondary outcomes will be collected by the study team from the patient chart and accompanying records and through patient interview. Continuous variables will be analyzed using t-tests and categorical variables will be analyzed using chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years
* Undergoing major urological surgery
* Consent to a rectus sheath blockade as part of their postoperative management

Exclusion Criteria:

* Patients under 18 years
* Local or systemic infection
* Patients who refuse consent
* Opioid tolerance
* History of chronic pain
* Psychiatric illness
* Allergy to local anesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Opioid requirement in first 24 hours after surgery | 24 hours
  Opioid requirement in first 24 hours after surgery

SECONDARY OUTCOMES:
Intra-operative opioid requirement | 3 - 6 hours
  Surgery times vary but on average the procedure being investigated takes 3 - 6 hours. Opioid administered during this time by the intra-operative anesthesiologist will be recorded for the study.
(Numerical Rating Scale) NRS pain score at 24 and 48 hours | 48 hours
  The NRS pain scale is a used to measure pain intensity. Patients are asked to rate their pain between 0 (no pain) and 10 (worst pain possible)
Severity of Nausea | 48 hours
  Rated as mild, moderate or severe by the patient
Number of vomiting episodes | 48 hours
  Number of discrete vomiting episodes per 24 hour period
Use of anti-emetics | 48 hours
  Name and total dose of anti-emetic per 24 hour period
Sedation score | 48 hours
  Patients will be rated as alert, drowsy, light sedation i.e. awakens with eye contact), moderate sedation (wakens to voice), deep sedation (wakes to physical stimulation but not to voice) and unrousable (no response to voice or physical stimulation).
Time to first bowel movement | Up to 7 days
  Time from end of surgery to first bowel movement.
Time to first mobilization | 48 hours
  Time from end of surgery to sitting on chair by bed
Duration of hospital stay | 7 - 14 days
  Time from end of surgery to ready for discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsui BC, Green JS, Ip VH. Ultrasound-guided rectus sheath catheter placement. Anaesthesia. 2014 Oct;69(10):1174-5. doi: 10.1111/anae.12849. No abstract available. PMID 25204242
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Siddiqui MR, Sajid MS, Uncles DR, Cheek L, Baig MK. A meta-analysis on the clinical effectiveness of transversus abdominis plane block. J Clin Anesth. 2011 Feb;23(1):7-14. doi: 10.1016/j.jclinane.2010.05.008. PMID 21296242
- [Background] Dutton TJ, McGrath JS, Daugherty MO. Use of rectus sheath catheters for pain relief in patients undergoing major pelvic urological surgery. BJU Int. 2014 Feb;113(2):246-53. doi: 10.1111/bju.12316. Epub 2013 Aug 13. PMID 23937574
- [Background] Tudor EC, Yang W, Brown R, Mackey PM. Rectus sheath catheters provide equivalent analgesia to epidurals following laparotomy for colorectal surgery. Ann R Coll Surg Engl. 2015 Oct;97(7):530-3. doi: 10.1308/rcsann.2015.0018. PMID 26414363